CLINICAL TRIAL: NCT03807076
Title: Modulating the Glucose-dependent Insulinotropic Polypeptide (GIP) System in Patients With Acromegaly Due to a Pituitary Tumor
Brief Title: Modulating the GIP System in Patients With Acromegaly Due to a Pituitary Tumor
Acronym: GA-9
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other); Aarhus University Hospital (Other); Aalborg University Hospital (Other); Odense University Hospital (Other); Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Mette Høy Jensen, Industrial PhD student, University of Copenhagen
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Acromegaly GA-9
Record Dates: First submitted 2019-01-15; First posted 2019-01-16 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Acromegaly Due to Pituitary Adenoma
MeSH Terms: conditions — Growth Hormone-Secreting Pituitary Adenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GIP-A (Other): Infusion of GIP-A alone as a study tool.
  Interventions: Other: GIP-A
- Placebo (Placebo Comparator): Saline
  Interventions: Other: Placebo

INTERVENTIONS:
Other: GIP-A — GIP-A
  Arms: GIP-A
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Modulation of the GIP System in Patients With Acromegaly Due to a Pituitary adenoma

DETAILED DESCRIPTION:
Aim: To determine the importance of the GIP system in patients with acromegaly who has paradoxical growth hormone secretion during an oral glucose tolerance test (OGTT) using a GIP antagonist (GIP-A).

Thirty participants (age 18-75 years) with normal kidney and liver parameters and hemoglobin levels will be included in a placebo-controlled cross-over study. The study consists of two study days with concomitant infusions of A) GIP-A or B) saline (placebo).

A paradoxical growth hormone secretion to an OGTT is here defined as an increase in plasma growth hormone levels of ≥30% from baseline based on a mean value of the definitions in the literature.

Regazzo et al. (2017) European Journal of Endocrinology 176, 543-553 Mukai et al. (2018) The Journal of Clinical Endocrinology and Metabolism 104(5), 1637-1644 Hage et al. (2019) The Journal of Clinical Endocrinology and Metabolism 104(5), 1777-1787 Scaroni et al. (2019) J Clin Endocrinol Metab 104(3), 856-862

ELIGIBILITY:
Inclusion Criteria:

* Patients under clinical investigation of acromegaly disease with normal kidney function, liver function and hemoglobin levels.

Exclusion Criteria:

* Medication for acromegaly, adenectomy, liver disease, uncontrolled anemia, severe heart disease, uncontrolled high blood pressure (>170/100 mmHg), current pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Growth hormone levels | 240 min
  Plasma growth hormone area under the curve (AUC)

SECONDARY OUTCOMES:
Glucose levels | 240 min
  Plasma glucose AUC
GIP levels | 240 min
  Plasma GIP AUC
Insulin levels | 240 min
  Serum insulin AUC
C-peptide levels | 240 min
  Serum C-peptide AUC
Insulin-like growth factor-1 (IGF-1) levels | 240 min
  Plasma IGF-1 AUC
Free fatty acids (FFA) levels | 240 min
  serum FFA AUC
Glucagon levels | 240 min
  plasma glucagon AUC
Ghrelin levels | 240 min
  plasma ghrelin AUC
GLP-1 levels | 240 min
  Plasma GLP-1 AUC
GLP-2 levels | 240 min
  Plasma GLP-2 AUC
Plasma cholesterol | 240 min
  Plasma cholesterol AUC
Plasma triglyceride | 240 min
  Plasma triglyceride AUC
Plasma TSH | 240 min
  Plasma TSH AUC
Plasma prolactin | 240 min
  Plasma prolactin AUC

CONTACTS AND LOCATIONS:
Overall Officials: Mette H Jensen, MSc, Principal Investigator — Department of Biomedical Sciences
Locations (1):
- Department of Biomedical Sciences, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No